CLINICAL TRIAL: NCT02403570
Title: Rotating Frame Relaxation Imaging in Patients With Multiple Sclerosis
Acronym: ROMUS
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Hannu Aronen, Professor, Turku University Hospital
Other Study IDs: T125/2014
Record Dates: First submitted 2015-03-10; First posted 2015-03-31 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive
Keywords: Multiple Sclerosis, MRI, rotating frame
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Multiple Sclerosis: Brain MRI using advanced MR techniques
  Interventions: Other: Brain MRI

INTERVENTIONS:
Other: Brain MRI

SUMMARY:
The aim of this study is to develop novel magnetic resonance imaging (MRI) protocols suitable for patients with multiple sclerosis using advanced MRI such as rotating frame relaxation imaging. In addition, the investigators want to study the correlation between advanced MRI parameters and clinical disease progression.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of relapsing remitting MS made according to the Poser, McDonald's or revised McDonald's criteria (Group I) before participating in the study
* Initial MS diagnosis of relapsing remitting form of the disease according to the criteria as mentioned above, and conversion into the secondary progressive phase of the disease as evaluated by the referring neurologist according to the clinical evaluation and confirmed by the study physician (Group II).
* Mental status: Patients must be able to understand the meaning of the study
* Informed consent: The patient must sign the appropriate Ethical Committee (EC) approved informed consent documents in the presence of the designated staff

Exclusion Criteria:

* Any other autoimmune disease than MS requiring immunomodulatory or immunosuppressive medication
* High-dose corticosteroid treatment within 30 days before participating in the study
* Prior medical history: Patient must have no history of serious cardiovascular, liver or kidney disease
* Any psychiatric condition that compromises the subject's ability to participate in the study
* Infections: Patient must not have an uncontrolled serious infection
* No contraindications for MRI (cardiac pacemaker, intracranial clips etc)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MS patients with relapsing-remitting or secondary progressive MS will be recruited from amongst the MS patients in the neurological outpatient policlinics in the Hospital District of Southwestern Finland.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2015-02; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
MR relaxation values 0 | Baseline
  Aim is to measure different quantitative MR relaxation values (e.g. Traff, T1rho) in different brain areas of patients with MS at baseline
MR relaxation values 1 | One year
  Aim is to measure different quantitative MR relaxation values (e.g. Traff, T1rho) in different brain areas of patients with MS after one year follow-up

SECONDARY OUTCOMES:
MR relaxation values and clinical markers 0 | Baseline
  Aim is to study the correlation between MR relaxation values and clinical markers of MS at baseline
MR relaxation values and clinical markers 1 | One year
  Aim is to study the correlation between MR relaxation values and clinical markers of MS after one year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Hannu Aronen, M.D., Ph.D., Principal Investigator — Turku University Hospital, Department of Diagnostic Radiology
Locations (1):
- Division of Clinical Neurosciences, Turku University Hospital, Turku, Finland